CLINICAL TRIAL: NCT02393872
Title: Developing and Implementing a Community-based Intervention to Create a More Supportive Social and Physical Environment for Lifestyle Changes to Prevent Diabetes in Vulnerable Families Across Europe.
Brief Title: Feel4Diabetes-study
Acronym: Feel4Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); University Ghent (Other); Technische Universität Dresden (Other); National and Kapodistrian University of Athens (Other); International Diabetes Federation (Other); Universidad de Zaragoza (Other); Medical University of Varna (Other); University of Debrecen (Other); Extensive Life Oy (Unknown)
Responsible Party: Principal Investigator, Yannis Manios, Associate Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 643708
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Prevention
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-risk families component (Experimental): School-based intervention and counselling sessions.
  Interventions: Behavioral: Feel4Diabetes-intervention
- All-families component (Experimental): School-based intervention.
  Interventions: Behavioral: Feel4Diabetes-intervention
- Control (No Intervention): Control group.

INTERVENTIONS:
Behavioral: Feel4Diabetes-intervention — Community-based intervention.
  Arms: All-families component; High-risk families component

SUMMARY:
The aim of the Feel4Diabetes-study is to develop, implement and evaluate a community-based intervention aiming to create a more supportive social and physical environment to promote lifestyle and behaviour change to prevent type 2 diabetes among families from low and middle income countries and from vulnerable groups in high income countries in Europe.

DETAILED DESCRIPTION:
The aim of the Feel4Diabetes-study is to develop, implement and evaluate a community-based intervention aiming to create a more supportive social and physical environment to promote lifestyle and behaviour change to prevent type 2 diabetes among families from low and middle income countries and from vulnerable groups in high income countries in Europe.

The Feel4Diabetes-intervention will be developed according to the results of systematic literature reviews, narrative reviews and surveys regarding existing research programs, legislation and policies as well as infrastructures, facilities and human resources, which will be conducted during the first phase of the project. It will be implemented in six Eurepean countries, namely Belgium, Bulgaria, Finland, Greece, Hungary and Spain. The process, impact, outcome, cost-effectiveness and scalability of the Feel4Diabetes-intervention will be evaluated and the results of the study will be disseminated via various communication channels.

ELIGIBILITY:
Inclusion Criteria:

* For children and their parents: low socioeconomic areas and/or vulnerable subgroups of population
* For children: first two grades of compulsory education.

Exclusion Criteria:

* Age range not within the inclusion criteria.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Harokopio University of Athens, Kallithea, Attica, Greece

REFERENCES:
- [Derived] Mahmood L, Moreno LA, Schwarz P, Annemans L, Cardon G, Hilal S, Rurik I, Iotova V, Usheva N, Tankova T, Anastasiou C, Manios Y, Gonzalez-Gil EM; Feel4Diabetes-Study Group. Socioeconomic Vulnerability and Its Associations With Dietary Patterns and Obesity Degree Among Children in Families Across Six European Countries: The Feel4Diabetes-Study. Pediatr Obes. 2026 Jan;21(1):e70072. doi: 10.1111/ijpo.70072. PMID 41558509
- [Derived] Mahmood L, Moreno LA, Schwarz P, Willems R, Cardon G, Hilal S, Rurik I, Iotova V, Bazdarska Y, Dimova R, Anastasiou K, Manios Y, Gonzalez-Gil EM; Feel4Diabetes-Study Group. A snapshot of country-specific dietary habits and obesity in European children: the Feel4Diabetes study. Eur J Pediatr. 2025 Feb 27;184(3):214. doi: 10.1007/s00431-025-06037-4. PMID 40016587
- [Derived] Cardon G, Chastin S, Van Stappen V, Huys N, Stefanova T, Chakarova N, Kivela J, Alberto Moreno L, Sandor Istvanne R, Androutsos O, Manios Y, De Craemer M. The Feel4Diabetes intervention: effectiveness on 24-hour physical behaviour composition in families at risk for diabetes development. Health Promot Int. 2022 Oct 1;37(5):daac092. doi: 10.1093/heapro/daac092. PMID 36287523
- [Derived] Kontochristopoulou AM, Karatzi K, Karaglani E, Cardon G, Kivela J, Wikstrom K, Iotova V, Tsochev K, Tankova T, Rurik I, Radone AS, Liatis S, Makrilakis K, Moreno LA, Manios Y. Sociodemographic, anthropometric, and lifestyle correlates of prediabetes and type 2 diabetes in europe: The Feel4Diabetes study. Nutr Metab Cardiovasc Dis. 2022 Aug;32(8):1851-1862. doi: 10.1016/j.numecd.2022.03.021. Epub 2022 Apr 2. PMID 35610084
- [Derived] Mahmood L, Gonzalez-Gil EM, Schwarz P, Herrmann S, Karaglani E, Cardon G, De Vylder F, Willems R, Makrilakis K, Liatis S, Iotova V, Tsochev K, Tankova T, Rurik I, Rado S, Moreno LA, Manios Y; Feel4Diabetes-Study Group. Frequency of family meals and food consumption in families at high risk of type 2 diabetes: the Feel4Diabetes-study. Eur J Pediatr. 2022 Jun;181(6):2523-2534. doi: 10.1007/s00431-022-04445-4. Epub 2022 Mar 30. PMID 35353229
- [Derived] Willems R, Tsoutsoulopoulou K, Brondeel R, Cardon G, Makrilakis K, Liatis S, Lindstrom J, Kivela J, Gonzalez-Gil EM, Gimenez-Legarre N, Usheva N, Iotova V, Tankova T, Antal E, Rurik I, Timpel P, Schwarz PEH, Manios Y, Annemans L. Cost-effectiveness analysis of a school- and community-based intervention to promote a healthy lifestyle and prevent type 2 diabetes in vulnerable families across Europe: the Feel4Diabetes-study. Prev Med. 2021 Dec;153:106722. doi: 10.1016/j.ypmed.2021.106722. Epub 2021 Jul 14. PMID 34271077
- [Derived] Huys N, Van Stappen V, Shadid S, De Craemer M, Androutsos O, Wikstrom K, Makrilakis K, Moreno LA, Iotova V, Tankova T, Nanasi A, Manios Y, Cardon G; Feel4Diabetes-study group. Effectiveness of a family-, school- and community-based intervention on physical activity and its correlates in Belgian families with an increased risk for type 2 diabetes mellitus: the Feel4Diabetes-study. BMC Public Health. 2020 Aug 12;20(1):1231. doi: 10.1186/s12889-020-09336-7. PMID 32787943
- [Derived] Manios Y, Lambrinou CP, Mavrogianni C, Cardon G, Lindstrom J, Iotova V, Tankova T, Rurik I, Stappen VV, Kivela J, Mateo-Gallego R, Moreno LAlpha, Makrilakis K, Androutsos O. Lifestyle Changes Observed among Adults Participating in a Family- and Community-Based Intervention for Diabetes Prevention in Europe: The 1st Year Results of the Feel4Diabetes-Study. Nutrients. 2020 Jun 30;12(7):1949. doi: 10.3390/nu12071949. PMID 32629949
- [Derived] Virtanen E, Kivela J, Wikstrom K, Lambrinou CP, De Miguel-Etayo P, Huys N, Vrauko-Toth K, Moreno LA, Usheva N, Chakarova N, Rado SA, Iotova V, Makrilakis K, Cardon G, Liatis S, Manios Y, Lindstrom J; Feel4Diabetes research group. Feel4Diabetes healthy diet score: development and evaluation of clinical validity. BMC Endocr Disord. 2020 May 6;20(Suppl 2):46. doi: 10.1186/s12902-020-0521-x. PMID 32370805
- [Derived] Androutsos O, Anastasiou C, Lambrinou CP, Mavrogianni C, Cardon G, Van Stappen V, Kivela J, Wikstrom K, Moreno LA, Iotova V, Tsochev K, Chakarova N, Ungvari T, Jancso Z, Makrilakis K, Manios Y; Feel4diabetes-study group. Intra- and inter- observer reliability of anthropometric measurements and blood pressure in primary schoolchildren and adults: the Feel4Diabetes-study. BMC Endocr Disord. 2020 Mar 12;20(Suppl 1):27. doi: 10.1186/s12902-020-0501-1. PMID 32164691
- [Derived] Kivela J, Wikstrom K, Virtanen E, Georgoulis M, Cardon G, Civeira F, Iotova V, Karuranga E, Ko W, Liatis S, Makrilakis K, Manios Y, Mateo-Gallego R, Nanasi A, Rurik I, Tankova T, Tsochev K, Van Stappen V, Lindstrom J; Feel4Diabetes research group. Obtaining evidence base for the development of Feel4Diabetes intervention to prevent type 2 diabetes - a narrative literature review. BMC Endocr Disord. 2020 Mar 12;20(Suppl 1):140. doi: 10.1186/s12902-019-0468-y. PMID 32164690
- [Derived] Manios Y, Mavrogianni C, Lambrinou CP, Cardon G, Lindstrom J, Iotova V, Tankova T, Civeira F, Kivela J, Jancso Z, Shadid S, Tsochev K, Mateo-Gallego R, Rado S, Dafoulas G, Makrilakis K, Androutsos O; Feel4Diabetes-study group. Two-stage, school and community-based population screening successfully identifies individuals and families at high-risk for type 2 diabetes: the Feel4Diabetes-study. BMC Endocr Disord. 2020 Mar 12;20(Suppl 1):12. doi: 10.1186/s12902-019-0478-9. PMID 32164646
- [Derived] Huys N, Van Stappen V, Shadid S, De Craemer M, Androutsos O, Lindstrom J, Makrilakis K, de Sabata MS, Moreno L, De Miguel-Etayo P, Iotova V, Rurik I, Manios Y, Cardon G; Feel4Diabetes-Study Group. Influence of Educational Level on Psychosocial Correlates and Perceived Environmental Correlates of Physical Activity in Adults at Risk for Type 2 Diabetes: The Feel4Diabetes-Study. J Phys Act Health. 2019 Dec 1;16(12):1105-1112. doi: 10.1123/jpah.2019-0003. Epub 2019 Oct 31. PMID 31672925